CLINICAL TRIAL: NCT04159480
Title: Facilitating Assessment of At-Risk Sailors Using Technology
Acronym: FAAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other); Military Suicide Research Consortium (Other)
Responsible Party: Principal Investigator, Lisa Brenner, Investigator, VA Eastern Colorado Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-2844
Record Dates: First submitted 2019-10-30; First posted 2019-11-12 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Psychological Distress

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes measures will be collected electronically
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Experimental - Cogito Companion (Experimental): Those allocated to Experimental arm will have access the Cogito Companion for a three-month period post-consent. Passive data collection will also occur during this period. As a secure, privacy-compliant mobile app, the Cogito Companion facilitates the non-invasive collection, transfer, integration, analysis, and reporting of objective behavioral indicators. The Cogito mobile sensing platform passively gathers behavioral information through an individual's normal smartphone usage. Measurements of location, call, and text patterns are recorded.
  Interventions: Device: Experimental - Cogito Companion
- Active Control (Active Comparator): Participants randomized to the Active Control group will download MyCAP and have access to resources housed within this app for a three-month period post-consent. Participants will be provided information regarding the mHealth Tool apps, and provided basic information on how to download the apps. As noted above, participants will be provided biweekly surveys .
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Device: Experimental - Cogito Companion — Cogito Companion
  Arms: Experimental - Cogito Companion
Behavioral: Active Control — Use of MyCAP
  Arms: Active Control

SUMMARY:
Randomized clinical trial with individuals being allocated to experimental (Cogito Companion) or Active Control arms. Those in the latter will receive information regarding widely available mobile self-help apps via a custom mobile app built in MyCAP. This same platform will be used to collect data regarding symptoms. Randomization will be stratified by gender, force (Surface, Aviation), and smartphone model (Android, I-Phone), as Cogito algorithms differ based on smartphone platforms. Participants will be willing Naval personnel being redeployed to CONUS. Data is also being collected (feasibility/acceptability) to inform future implementation..

ELIGIBILITY:
Inclusion Criteria.

* Member of the Navel Surface or Aviation Forces;
* Age: 18-55 years at the time of enrollment;
* Ability to provide verbal and electronic informed consents;
* Ownership of smartphone;
* Willingness to use smartphone and personal data plan to participate.

Exclusion Criteria.

* Having redeployed (returning to the Continental United States) more than twelve months (approximately) prior to consent.
* Having an iPhone (until later in 2019 when the Cogito Corporation plans to release the iOS version of the Cogito Companion app).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brenner, Ph.D., Principal Investigator — VA/University of Colorado
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 279 Naval personnel were enrolled and randomized - 139 participants to Cognito Companion and 140 to Active Control
Units Other Than Participants: Online Assessment
Period: Overall Study
Arm/Group | Experimental - Cogito Companion | Active Control
Started | 139; 139 Online Assessment | 140; 140 Online Assessment
Completed | 139; 139 Online Assessment | 140; 140 Online Assessment
Not Completed | 0; 0 Online Assessment | 0; 0 Online Assessment

BASELINE CHARACTERISTICS:
Population: Randomized
Groups:
- Cogito: Randomized to Cogito
- Active Control: Randomized to Control
- Total: Total of all reporting groups
Arm/Group | Cogito | Active Control | Total
Number analyzed (Participants) | 139 | 140 | 279
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (6.8) | 28.3 (6.7) | 28.5 (6.8)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender of Participants Population: Evaluated characteristic by group
  Participants
    Gender: Male | 109 | 109 | 218
    Gender: Female | 28 | 28 | 56
    Gender: Declined | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian/White | 89 | 82 | 171
  Race/Ethnicity: Black/African American | 26 | 22 | 48
  Race/Ethnicity: Native American/Alaskan | 3 | 1 | 4
  Race/Ethnicity: Asian | 7 | 11 | 18
  Race/Ethnicity: Pacific Islander | 1 | 0 | 1
  Race/Ethnicity: Other | 2 | 9 | 11
  Race/Ethnicity: Multiple Races | 8 | 9 | 17
  Race/Ethnicity: Declined to Answer | 3 | 6 | 9
Ranomized to Cogito or Active Control [Count of Participants; unit: Participants] | 139 | 140 | 279

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Cogito Participants Reported Being Satisfied
Description: To measure the percentage of participants randomized to Cogito who were satisfied, a 'Client Satisfaction Questionnaire' was distributed to participants to complete and return. Responses were collected and evaluated to find the percentage of participant satisfaction.
Time Frame: From Baseline to Follow-Up, Approximately 3 months
Population: Participant Satisfaction
Measure: Number; unit: percentage of participants
Arm/Group | Cogito
Number analyzed (Participants) | 40
percentage of participants | 52

ADVERSE EVENTS:
Time Frame: From Baseline to Follow-Up, Approximately 3 Months
Description: All cause death and serious adverse event related to study participation
Groups:
- Cogito: Adverse events for Cogito group.
- Active Control: Adverse events for Active Control group.
Arm/Group | Cogito | Active Control
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/140
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/140
Other Adverse Events (participants affected / at risk) | 0/139 | 0/140

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT04159480/Prot_002.pdf
  • Statistical Analysis Plan (2023-05-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT04159480/SAP_003.pdf